CLINICAL TRIAL: NCT02116322
Title: EUS-guided Fine Needle Tissue Acquisition of Solid Pancreatic Mass Lesions Using a Novel Corkscrew Technique: a Pilot Study
Brief Title: Endoscopic Ultrasound (EUS) Guided Fine Needle Aspiration (FNA) EUS-FNA of Solid Pancreatic Mass Lesions Using a Novel Corkscrew Technique: a Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study stopped as the used needle was difficult to maneuver in the corkscrew method being studied so no more participants were included.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00090101
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pancreatic mass (Experimental): Patients with pancreatic mass presenting for EUS-FNA
  Interventions: Procedure: EUS-FNA with Corkscrew technique; Device: Expect 19 G Flex needle

INTERVENTIONS:
Procedure: EUS-FNA with Corkscrew technique
Device: Expect 19 G Flex needle
  Other Names: Expect 19G Flex needle; Boston scientific

SUMMARY:
This research is being done to investigate if a new technique to biopsy the pancreas will lead to a larger amount tissue material that can be analyzed. Investigators have called the technique the "corkscrew" technique and believe it will allow obtaining a larger biopsy sample during the endoscopic ultrasound examination. The corkscrew technique uses a clockwise rotational movement to drive the needle into the pancreatic mass (like a wine bottle opener twists and buries itself into a cork). It is believed that this will lead to a better biopsy sample than the usual way and therefore result in a higher chance of a diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* In-patients and out-patients between the age of 18 and 90 years with solid pancreatic masses presenting for EUS-Fine Needle Aspiration (FNTA)

Exclusion Criteria:

* Uncorrectable coagulopathy (INR > 1.5)
* Uncorrectable thrombocytopenia (platelet < 50,000)
* Uncooperative patients
* Pregnant women (women of childbearing age will undergo urine pregnancy testing, which is routine for all endoscopic procedures)
* Refusal to consent form
* Prior negative FNTA
* In situ metallic biliary stents
* Predominantly cystic lesions
* Inaccessible lesions to EUS

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mouen A Khashab, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between 7/18/14 and 2/18/15 in an academic tertiary center
Pre-assignment Details: A total of 4 participants were enrolled. However, 3 participants were excluded before being assigned to the study arm because the performing endoscopist didn't find it possible to do the procedure due to the unfavorable size of the mass or technical difficulty.
Groups:
- Pancreatic Mass: Patients with pancreatic mass presenting for EUS-FNA
  EUS-FNA with Corkscrew technique
  Expect 19 G Flex needle
Period: Overall Study
Arm/Group | Pancreatic Mass
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pancreatic Mass
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 80
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Pancreatic Mass
Number analyzed (Participants) | 1
participants | 0

2. Secondary Outcome: Diagnostic Yield of the FNA Using Corkscrew Technique
Description: Diagnostic yield was defined as the proportion of masses in which the amount of FNA-obtained cellular material was enough for the histopathologist to make the pathological diagnosis.
Time Frame: 30 days
Measure: Number; unit: percentage of masses
Arm/Group | Pancreatic Mass
Number analyzed (Participants) | 1
percentage of masses | 0

ADVERSE EVENTS:
Arm/Group | Pancreatic Mass
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes